CLINICAL TRIAL: NCT00242554
Title: Open-label Phase IV Clinical Trial to Evaluate the Safety and Tolerability of Zoledronic Acid in Patients With Prostate Cancer and Bone Metastases
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CZOL446EMX01
Record Dates: First submitted 2005-10-09; First posted 2005-10-20 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Bone Metastases; Zoledronic acid
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Zoledronic Acid

INTERVENTIONS:
Drug: Zoledronic acid

SUMMARY:
To assess the effects of i.v. zoledronic acid 4 mg with respect to safety and tolerability

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histological confirmed diagnosis of carcinoma of the prostate
* Current or previous evidence of metastatic disease to the bone
* Receiving currently or not, hormonal therapy
* ECOG performance status of 0, 1, or 2

Exclusion Criteria:

* Patients with abnormal renal function as evidenced by either a serum creatinine determination 1.5 x or greater above the upper limit of normal, or by a calculated creatinine clearance of 60 ml/minute or less.
* Corrected serum calcium concentration, adjusted for serum albumin < 8.0 mg/dl (2.00 mmol/L).
* WBC<3.0x10^9, ANC < 1500/mm3, Hb < 8.0 g/dL, platelets < 75 x 10^9/L.
* Liver function tests >2.5 ULN, serum creatinine >1.5 ULN.
* Patients with another non malignant disease, which could confound the evaluation of primary endpoints, or prevent the patient complying with the protocol.
* Known hypersensitivity to zoledronic acid or other bisphosphonates or each of the compounds which perform the formula.

Other protocol-related inclusion / exclusion criteria may apply

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2002-10; Primary Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the tolerability and safey of zoledronic acid 4mg, IV, for the following eficacy metrics: QoL, Safety (Aes) and evaluation of pain

SECONDARY OUTCOMES:
No secondary outcomes/objectives planned

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals